CLINICAL TRIAL: NCT05795972
Title: Efficacy Evaluation of Inulin Supplementation on Metabolic Control and Akkermansia Muciniphila Levels in Patients With Type 1 Diabetes: a Pilot Study
Brief Title: Inulin Supplementation in Patients With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, OJETTI VERONICA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3099
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Inulin; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inulin supplementation (Experimental)
  Interventions: Dietary Supplement: inulin
- standard therapy (Active Comparator)
  Interventions: Other: standard therapy

INTERVENTIONS:
Dietary Supplement: inulin — patients treated with standard therapy with a supplementation of Inulin 6g twice a day for 3 months.
  Arms: inulin supplementation
Other: standard therapy — control group (patients treated also with standard therapy)
  Arms: standard therapy

SUMMARY:
The aim of this study is to compare the glycemic and metabolic control of type 1 diabetic patients in replacement therapy with insulin, comparing those treated with a supplementation of prebiotics (inulin) and those treated with a placebo.

Therefore, the primary objective of the study is represented by the proportion of patients with better glycemic control (basal and post-prandial euglycemia time) and optimal metabolic control (HbA1c, lipid profile, C-RP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with T1D, diagnosed before 35 years of age will be enrolled

Exclusion Criteria:

* advanced complications of T1D (established renal failure, severe retinopathy and diabetic neuropathy)
* BMI> 30 kg / m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
glycemic control | 3 months
  represented by the proportion of patients with better glycemic control (basal and post-prandial euglycemia time) and optimal metabolic control (HbA1c, lipid profile, C-RP).

SECONDARY OUTCOMES:
akkermania levels | 3 months
  evaluate the presence of Akkermansia in the gut microbiota at enrollment, and to compare its quantitative modification from the beginning to the end of the therapy, comparing inulin vs a control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy